CLINICAL TRIAL: NCT06421103
Title: Investigating Micro-dosing of Indocyanine Green (ICG) for Intraoperative Perfusion Assessment in Children.
Brief Title: Micro-dosing Indocyanine Green (ICG) in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 23BO01
Record Dates: First submitted 2024-01-08; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Perfusion; Fluorescence Imaging; Gastrointestinal Tract Disorders; Genitourinary Disease
Keywords: Paediatric Surgery; Pediatric Surgery; Fluorescence; Imaging; Fluorescence Guided Surgery (FGS); Intra-operative perfusion assessment; Indocyanine Green
MeSH Terms: conditions — Digestive System Diseases; Urogenital Diseases | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: Dose escalation with backfilling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Micro-dosing Indocyanine Green (ICG) (Experimental): Multiple dose levels of intravenous Indocyanine Green (ICG) administered intra-operatively. Starting dose will be 10% of standard (for the study institution) and escalated as per protocol.
  Interventions: Drug: Indocyanine Green (ICG)

INTERVENTIONS:
Drug: Indocyanine Green (ICG) — Cohorts will receive 0.01 mg/kg, 0.02 mg/kg, 0.04mg/kg, 0.06 mg/kg, or 0.08 mg/kg intra-venous ICG at surgery. Patients will be consecutively allocated to different doses as per protocol.
  Other Names: Verdye by DiagnosticGreen

SUMMARY:
The goal of this cohort study is to identify the lowest dose of Indocyanine Green (ICG) that achieves satisfactory intra-operative fluorescence for the assessment of gastrointestinal or genitourinary tract perfusion in children.

DETAILED DESCRIPTION:
Indocyanine Green (ICG) fluorescence-guided surgery (FGS) can be used to assess gastrointestinal and genitourinary tract perfusion intra-operatively. In adults, the use of ICG has been shown to improve surgical outcomes. ICG is safely used intra-operatively in children, but there is a lack of evidence regarding the lowest clinically useful dose of ICG.

This is a single centre open-label dose escalation study that aims to:

1. identify the minimal clinically useful dose of ICG for intra-operative perfusion assessment in children (0 - 18 years old)
2. assess the safety profile of intra-operative ICG in children
3. characterise the intra-operative fluorescence of ICG in children

ELIGIBILITY:
Inclusion Criteria:

* Children aged ≤18 years of age
* Elective surgery including gastrointestinal or genitourinary tract perfusion assessment

Exclusion Criteria:

* Renal and liver dysfunction
* Active infection
* Coagulopathy
* Complex congenital heart defect
* Previous documented allergy to ICG injection or other iodinated contrast agents
* Patients suffering from hyperthyroidism or autonomic thyroid adenomas
* Premature infants or neonates in whom exchange transfusion is indicated, due to the hyperbilirubinaemia risk
* Concurrent use of sodium bisulphite-containing preparations, such as certain heparin preparations

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Minimum clinically useful dose of ICG in children | 60 minutes (intra-operative)
  Identify the minimum dose of ICG at which intra-operative perfusion assessment is achieveable. Assessment will be based objectively on mean fluorescence intensity and the fluorescence-time curve, and subjectively by the operating surgeon.
Number of adverse drug events at each dose level | 30 days
  An appreciably harmful or unpleasant reaction, resulting from an intervention related to the use of a medicinal product, which predicts hazard from future administration and warrants prevention or specific treatment, or alteration of the dosage regimen, or withdrawal of the product

SECONDARY OUTCOMES:
Surgical complications | 30 days
  Intra-operative and early postoperative complications and mortality (defined as an event observed within 30 days after surgery). Frequency and details.
Post-operative morbidity | 90 days
  Further procedures, complications and mortality occuring within the 30 - 90 day time period (late post-operative complications). Frequency and details.
Length of stay | 90 days
  Time in hospital post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Giuliani, Principal Investigator — Great Ormond Street Hospital
Locations (1):
- Great Ormond Street Hospital for Children, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No